CLINICAL TRIAL: NCT06573099
Title: A Real-World Study on Extranodal Lymphoma
Status: Not yet recruiting | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, First Deputy Director, Hematology Department, Ruijin Hospital
Other Study IDs: EXPECT-02
Record Dates: First submitted 2024-08-08; First posted 2024-08-27 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Lymphoma; Lymphoma, B-Cell; Lymphoma, Non-Hodgkin; Extranodal Lymphoma; Diffuse Large B Cell Lymphoma
Keywords: LYMPHOMA; EXTRANODAL; DLBCL
MeSH Terms: conditions — Lymphoma; Lymphoma, B-Cell; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No interventions need to be specified for this study — No interventions need to be specified for this study

SUMMARY:
The aim of this study is to prospectively collect clinical information on patients with extranodal lymphoma, and to explore the best therapeutic strategies in the real-world population.

DETAILED DESCRIPTION:
Lymphoma is a common hematological malignancy. Many different pathologic types of lymphoma can originate in extranodal organs or be associated with extranodal organ involvement. For lymphoma with extranodal involvement, conventional regimens often cannot provide satisfactory results for patients. This study aims to prospectively collect clinical information on patients with extranodal DLBCL, including the distribution of involved sites, clinical and molecular characteristics of different lymphoma subtypes, clinical treatment protocols, and prognosis, to explore the the best therapeutic strategies in the real-world population.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years (including 18 years old).
2. Patients newly diagnosed with non-Hodgkin lymphoma with extranodal involvement, whether it is primary, secondary, or cannot be determined.
3. Patients who have received systematic clinical treatment.
4. Patients with measurable lesions, at least containing one effective evaluation of efficacy.

Exclusion Criteria:

1. Patients who only receive supportive treatment.
2. Patients who cannot obtain effective evaluation data of efficacy.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients with histologically confirmed diagnosis of non-Hodgkin lymphoma with extranodal involvement.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2029-09-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Baseline up to data cut-off (up to approximately 1 year)
  Progression-Free Survival (PFS) will be defined from the date of starting therapy and the date of disease progression, relapse or death from any cause.

SECONDARY OUTCOMES:
Overall Survival (OS) | Baseline up to data cut-off (up to approximately 1 year)
  Overall Survival (OS) will be defined from the start date of therapy to the date of death from any cause.

IPD SHARING:
Plan to Share IPD: Undecided